CLINICAL TRIAL: NCT01151566
Title: Can US With CEUS Replace the Nonenhanced CT Scan in Patients With Contraindication to CT Contrast Agent
Brief Title: Can Ultrasound Replace Computed Tomography (CT) Scan in Those Unable to Have Computed Tomography (CT) Contrast Agents
Acronym: CEUS_CT
Status: Completed | Type: Observational
Sponsor: Foothills Medical Centre (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Stephanie R Wilson, MD, Clinical Professor of Radiology University of Calgary, Foothills Medical Centre
Other Study IDs: 21982
Record Dates: First submitted 2010-06-08; First posted 2010-06-28 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Nephrotoxicity of CT Contrast Agents; CT Scans in Those With Renal Compromise; Sensitivity to CT Contrast Agents; US With CEUS as Replacement for Unenhanced CT Scan
Keywords: Ultrasound; Contrast enhanced Ultrasound (CEUS); Nephrotoxicity; CT contrast agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Renal Compromise: Those referred for CT scan with identified renal compromise necessitating use of no contrast agent
- Sensitivity to CT Contrast Agents: Those referred for CT scan with prior demonstration of contrast sensitivity requiring use of no contrast

SUMMARY:
Computed tomography (CT) scan, performed with contrast enhancement, is one of the most commonly requested examinations in diagnostic imaging. In a patient with an elevated creatinine or an allergy to contrast agents, the scan may be performed without the benefit of contrast enhancement. Ultrasound (US), performed with contrast agent enhancement does not have any nephrotoxicity and may be performed on patients with CT contrast allergy. The investigators propose that US with Contrast enhanced ultrasound (CEUS) is superior to unenhanced CT scan in this population.

DETAILED DESCRIPTION:
Contrast enhanced computed tomography (CT) is one of the most common investigations performed in any radiology department, used widely in evaluating pathology in any part of the body.

Historically, it is well known that the use of contrast agents for CT scans may result in nephropathy, or renal failure. Nephrotoxicity associated with the injection of CT contrast agents may occasionally occur in healthy individuals and more commonly in those with borderline renal function. If abnormal kidney function is known to exist in a patient sent for CT scan, the examination is performed without the valuable assistance of contrast enhancement. Further, if prior hypersensitivity to the contrast agent for CT scan is known, again, the scan will be performed without the use of contrast agent.

Ultrasound (US) performed conventionally in grayscale and with Doppler is able to evaluate most abdominal and pelvic organs and also provides vascular information related to large vessel blood flow. Contrast enhanced ultrasound (CEUS) provides more precise information on blood flow than is available with Doppler and has been shown to be comparable to CT scan in some circumstances. We believe that a comparison of conventional US, with CEUS, and unenhanced CT scan would clearly favor ultrasound for detection of soft tissue pathology on the basis of its inherent tissue contrast differentiation.

ELIGIBILITY:
Inclusion Criteria:

* unenhanced CT scan of abdomen
* known renal compromise
* known hypersensitivity to CT contrast agents

Exclusion Criteria:

* CT scan performed with contrast agent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for unenhanced CT scan on the basis of renal compromise of CT contrast agent sensitivity will be eligible for recruitment for our study.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Demonstration of superiority of US with CEUS over nonenhanced CT scan (NECT) for observations and interpretation of findings | January 31, 2011
  Superiority of US over nonenhanced CT scan will be shown in a blind read by independent interpretation of each study by two experienced radiologists. All positive observations and interpretations will be documented. A comparison will be performed against a truth panel based on a compilation of the patient's entire clinical record and outcome.
  We hypothesize CT will result in multiple indeterminate examinations, and that all solid organ pathology will be more optimally characterized on US with contrast enhancement than on CT. Multiple other observations will be equal between the two studies.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie R Wilson, MD, Principal Investigator — Clinical Professor University of Calgary
Locations (1):
- Diagnostic Imaging Foothills Medical Centre, Calgary, Alberta, Canada